CLINICAL TRIAL: NCT03095248
Title: Phase 2 Trial of Selumetinib in Patients With Neurofibromatosis Type II Related Tumors
Brief Title: Trial of Selumetinib in Patients With Neurofibromatosis Type II Related Tumors
Acronym: SEL-TH-1601
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results review of patient data
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL-TH-1601; 2016-8833 (Other: Institutional review board)
Record Dates: First submitted 2017-03-08; First posted 2017-03-29 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Neurofibromatosis 2; Vestibular Schwannoma; Meningioma; Ependymoma; Glioma
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Meningioma; Ependymoma; Glioma | interventions — AZD 6244

STUDY DESIGN:
Intervention Model Description: All participants with neurofibromatosis type 2 (NF2) will be stratified based upon tumor type. Vestibular schwannomas are assigned and analyzed as Stratum 1 and all other NF2 associated tumor types will be analyzed as Stratum 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum 1 - NF2 related vestibular schwannomas (Experimental): Stratum 1 included patients with NF2 with vestibular schwannomas who exhibit hearing loss. Participants received continuous twice daily dosing of selumetinib. Dosing was based on BSA calculated at the beginning of each course. One course is equivalent to 28 days. Therapy continued for up to two years (26 courses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selumetinib
- Stratum 2: other NF2 related tumors (meningiomas and ependymoma) (Experimental): Stratum 2 will include patients who have progressive lesions other than VS (including non-vestibular schwannomas, meningiomas, and spinal cord lesions). Participants will receive continuous twice daily dosing of selumentinib. Dosing is based on BSA calculated at the beginning of each course. One course is equivalent to 28 days. Therapy may continue for up to two years (26 courses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Continuous twice daily dosing; oral agent
  Other Names: AZD6244

SUMMARY:
In this research study the researchers want to learn more about the effects (both good and bad) the study drug selumetinib has on participants with neurofibromatosis type II (NF2) related tumor.

The researchers are asking patients with NF2 related tumors to be in the study, because their hearing has decreased and/or their NF2 related tumor has started to grow.

The goals of this study are:

* Determine if selumetinib will stop NF2 related tumors from growing
* Measure the changes in hearing after receiving selumetinib for 6 months.
* Determine if selumetinib improves how participants feel (physically and emotionally) and how participants can perform daily activities.
* Examine tumor tissue, if available, in a laboratory to see if NF2 related tumors have targets of selumetinib.

DETAILED DESCRIPTION:
This is a Phase 2 trial to assess the hearing response rate and radiographic response of VS in children and young adults with NF2 who are treated with selumetinib. Dosing will be based on BSA calculated at the beginning of each course.

Selumetinib is taken orally twice a day continuously. One course is equivalent to 28 days. Therapy may continue for up to two years (26 courses) in the absence of disease progression or unacceptable toxicity. Dose modifications will be based on Body Surface Area (BSA).

In December, 2022 the investigator closed the Stratum 1 arm. Stratum 2 is reserved for patients who exhibit growth of a tumor(s) besides vestibular schwannoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the NF2 gene.

The NIH criteria includes presence of:

* Bilateral vestibular schwannomas, OR
* First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity.

The Manchester criteria includes presence of:

* Bilateral vestibular schwannomas, OR
* First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
* Unilateral vestibular schwannoma AND any two of: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
* Multiple meningiomas (two or more) AND unilateral vestibular schwannoma OR any two of: schwannoma, glioma, neurofibroma, cataract.

  - Patients do not need to have a histologic diagnosis in order to start therapy but must have measurable disease (in 2 dimensions) on MRI scan to be eligible.
* For Stratum 1: Patients must have a target VS with the following qualities:
* Associated with a word recognition score of < 85% and > 0% AND
* Documented progression defined as: Either progressive hearing loss or progressive tumor growth in last 18 months defined as ≥ 20% increase in volume.
* For Stratum 2: Patients must not meet the eligibility criteria as stated for Stratum 1 and have a target lesion that has exhibited progression.
* Progression is defined as: ≥ 25% increase in sum of the products of perpendicular diameters of lesions in the preceding 18 months; any new lesion; or clinical deterioration related to disease.

  - Patients must be able to swallow capsules
  * Age:
* Patients must be ≥ 3 years to ≤ 45 years of age at start of treatment

  - Prior Therapy
* Since there is no standard effective chemotherapy for patients with NF2 and vestibular schwannomas, meningiomas, or ependymomas patients may be treated on this trial without having received prior medical therapy directed at their VS, meningiomas, or ependymomas.
* Since selumetinib is not expected to cause substantial myelosuppression, there will be no limit to number of prior myelosuppressive regimen for these NF2 patients.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, biologic therapy or radiotherapy prior to entering this study except for alopecia.
* Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks if nitrosourea.
* Biologic agent: Patient must have received their last dose of the biologic agent ≥ 7 days prior to study registration. For biologic agents that have a prolonged half-life, at least three half-lives must have elapsed prior to registration
* Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration

  - Corticosteroids:
* Patients who are receiving dexamethasone or other corticosteroids must be on a stable or decreasing dose for at least 1 week prior to registration. It is recommended that patients be off all steroid therapy or receive the least dose that will control their neurologic symptoms

  - Prior radiotherapy
* XRT: ≥ 6 months must have elapsed if prior XRT to vestibular schwannoma or other tumor.

  - Stem Cell Transplant or Rescue without TBI:
* No evidence of active graft vs. host disease and ≥ 3 months must have elapsed since transplant.

  - Performance Status:
* Karnofsky ≥ 60% for patients > 16 years of age
* Lansky ≥ 60 for patients ≤ 16 years of age.

  - Organ Function Requirements
* Adequate Bone Marrow Function Defined as:

  - Peripheral absolute neutrophil count (ANC) ≥ 1500/μL
* Platelet count ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to registration)
* Hemoglobin ≥ 9 g/dL (may receive RBC transfusions)
* Adequate Renal Function Defined as:
* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or
* A serum creatinine ≤1.5×ULN for age and sex
* Adequate Liver Function Defined as:
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
* AST(SGOT)/ALT(SGPT) ≤2.5×ULN institutional upper limit of normal for age
* Central Nervous System Function:

  - Patients with seizure disorder may be enrolled if they are receiving non-enzyme inducing anticonvulsants and the seizures are well controlled.
* Cardiac Function

Adequate cardiac function defined as:

* LVEF ≥55% by ECHO
* QTc interval ≤450 msecs by EKG
* Hypertension
* Patients, 3 to < 18 years of age must have a blood pressure that is ≤ 95th percentile for age, height and gender at the time of registration.
* Patients who are ≥18 years of age must have a blood pressure that is <140/90 mm of Hg at the time of registration.

Patients may be on blood pressure medication provided that it is not on the contraindicated list and that the medication has not been adjusted in the previous 3 months.

- Growth factors: All colony forming growth factor(s) have been discontinued for at least one week prior to registration (filgrastim, sargramostim, and erythropoietin). For patients on long acting growth factors, the interval should be two weeks.

* Inclusion of Women and Minorities Both males and females of all races and ethnic groups are eligible for this study.
* Informed Consent:

All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. The effects of selumetinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for four weeks after dosing with selumetinib ceases. The selumetinib manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle. Women of child-bearing potential must have a negative pregnancy test prior to study registration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Note: Female subjects are considered "of child-bearing potential" if they are anatomically and physiologically capable of becoming pregnant. For girls of normal reproductive potential, the possibility of becoming pregnant requires ovulatory menstrual cycles and heterosexual intercourse. Although the timing of ovulation relative to menarche is variable, there is consistent evidence that some girls may have ovulatory cycles prior to menarche, and that, in healthy populations, regular ovulation may begin within a few months of menarche. Therefore, menarche is the most feasible clinical indicator of the biological potential for pregnancy.

Male patients with sexual partners who are pregnant or who could become pregnant (i.e. women of child-bearing potential) must use acceptable, effective and reliable methods of contraception during the study and for at least 12 weeks after the last dose of selumetinib or for longer if required, depending on the prescribing information of the combination or concomitantly administered medications.

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) that is likely to interfere with the study procedures or results
* Patients who are currently receiving another investigational drug within 4 weeks prior to the first dose of study treatment, or within a period during which the investigational drug or systemic anticancer treatment has not been cleared from the body (e.g. a period of 5 'half-lives'), whichever is the most appropriate and as judged by the investigator are not eligible.
* Patients who have taken another BRAF inhibitor such as Vemurafenib or Dabrafenib prior to study registration are not eligible. Prior treatment with selumetinib or another MEK inhibitor is not allowed.
* Patients with QTc interval of > 450 msec
* Patients who require enzyme inducing anti-convulsants to control seizures.
* Anticoagulation: Patients receiving coumadin are eligible but must have their PT and INR monitored prior to each 4 week course.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
* The following cardiac conditions:

  a. Uncontrolled hypertension in adults (BP ≥ 140/90 mmHg despite medical therapy) b. Acute coronary syndrome within 6 months prior to starting treatment c. Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy (Appendix H) d. Symptomatic heart failure NYHA Class II-IV, prior or current cardiomyopathy, or severe valvular heart disease (Appendix I) e. Prior or current cardiomyopathy including but not limited to the following: i. Known hypertrophic cardiomyopathy ii. Known arrhythmogenic right ventricular cardiomyopathy

  f. Previous moderate or severe impairment of left ventricular systolic function (LVEF <45% on echocardiography or equivalent on MuGA) if known even if full recovery has occurred.

  g. Severe valvular heart disease h. Baseline Left ventricular ejection fraction (LVEF) below the LLN or <50% measured by echocardiography or institution's LLN for MUGA i. Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
* Ophthalmological conditions as follows:

  1. Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion
  2. Intraocular pressure (IOP) > 21 mmHg or uncontrolled glaucoma (irrespective of IOP)
* Major surgery within 4 weeks of starting selumetinib. Portacath insertion, G Tube placement, and insertion of ventriculoperitoneal shunt are not considered major surgeries.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib or combination medications or any excipient of these medicinal products.
* History of a medical or psychiatric illness, that in the investigator's judgment renders the patient incapable of further therapy on this protocol
* Patients with progressive disease associated with significant or disabling clinical symptoms requiring immediate intervention with surgery or radiation therapy are not eligible.

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trent Hummel, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cincinnati Children's Hospital Medical Center home page — https://www.cincinnatichildrens.org/service/c/cancer-blood

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified through referrals and from the PIs current patient population. All patients were enrolled at Cincinnati Children's Hospital Medical Center. The study was opened to enrollment on 05/08/2017 and closed to accrual on 06/09/2024,
Pre-assignment Details: There were a total of 10 participants consented who met eligibility criteria and received study interventions.
Period: Overall Study
Arm/Group | Stratum 1 - NF2 Related Vestibular Schwannomas | Stratum 2: Other NF2 Related Tumors (Meningiomas and Ependymoma)
Started | 1 | 9
Completed | 1 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There will be two treatment strata. Stratum 1 is for those patients who have a target vestibular schwannoma which is causing hearing loss. Stratum 2 will be reserved for patients who exhibit growth of a tumor(s) besides vestibular schwannoma and are therefore not eligible for stratum 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 - NF2 Related Vestibular Schwannomas | Stratum 2: Other NF2 Related Tumors (Meningiomas and Ependymoma) | Total
Number analyzed (Participants) | 1 | 9 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 8 | 9
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 1 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 0 | 6 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 6 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 9 | 10

OUTCOME MEASURES:

1. Primary Outcome: Stratum 1- Number of Patients With Hearing Response at 24 Weeks as Measured by Word Recognition
Description: The primary endpoint for the Stratum 1 is hearing response at 24 weeks, defined as an improvement in word recognition score above the 95% critical difference, taking as reference the baseline word recognition score. Audiology will include measurement of pure tone thresholds and determination of word recognition scores. Word recognition scores measure the ability to recognize (as opposed to detect) auditory information. Patients are presented a list of 50 words at a fully audible level and the percentage identified correctly is the score. This study will use full 50-item monosyllable lists and standardized recordings.
  This Outcome Measure was pre-specified to be assessed only within the Stratum 1 Arm/Group.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 - NF2 Related Vestibular Schwannomas
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Radiographic Tumor Response
Description: To determine the radiographic response rate for Stratum 1 and Stratum 2. Specifics for each stratum are defined in the Arms/ Groups.
Time Frame: Through study completion up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Stratum 1: NF2 Tumor (Vestibular Schwanomas): Response and progression for vestibular schwannomas will be evaluated in this study using the Response Evaluation in Neurofibromatosis and Schwannomatosis (REiNS) criteria. Response and progression for stratum 1 will not be evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) or by MacDonald Criteria, since they may underestimate progression in these irregularly shaped tumors. However, linear measurements utilizing RECIST will be collected as part of the trial for comparison with volumetric measurements. Linear measurements utilizing RECIST will be used for non-target lesions on stratum 1.
  REiNS criteria for target lesions:
  Radiographic Response (RR) At least a 20% decrease in the volume of the target lesions, taking as reference the baseline volume.
  Progressive Disease (PD) At least a 20% increase in the volume of the target lesion, taking as reference the lower volume during treatment Stable Disease (SD) Does not meet criteria for radiographic response or for progressive disease.
  Non-target lesions (RECIST criteria) Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level
  Incomplete Response/ Stable Disease (SD): Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits
  Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
- Stratum 2- NF2 Tumors (Non-vestibular Schwanoma (VS)): Stratum 2 Response and progression for non-VS tumor by MacDonald Criteria as measured by Complete responses, partial response, stable disease or progressive disease.
Arm/Group | Stratum 1: NF2 Tumor (Vestibular Schwanomas) | Stratum 2- NF2 Tumors (Non-vestibular Schwanoma (VS))
Number analyzed (Participants) | 1 | 9
Participants | 1 | 9

ADVERSE EVENTS:
Time Frame: Patients will be monitored for adverse events beginning on day 1 of study treatment and continue for the duration of time on study treatment, which may continue for up to 26 courses (approximately 2 years). Adverse events will also be monitored for 30 days post discontinuation of study treatment.
Description: Adverse Event Reporting Description for this study uses the same definitions in the link above.
Arm/Group | Stratum 1 - NF2 Related Vestibular Schwannomas | Stratum 2: Other NF2 Related Tumors (Meningiomas and Ependymoma)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/9
Other Adverse Events (participants affected / at risk) | 1/1 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 - NF2 Related Vestibular Schwannomas (N=1) | Stratum 2: Other NF2 Related Tumors (Meningiomas and Ependymoma) (N=9)
Grade 4 hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Grade 3 hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Grade 2 facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Grade 3 salivary gland infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 - NF2 Related Vestibular Schwannomas (N=1) | Stratum 2: Other NF2 Related Tumors (Meningiomas and Ependymoma) (N=9)
CPK increased (Investigations) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders-other: mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders-other: stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Localized Edema (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 6 (9)
Infections and Infestations-other: erythema toe (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-other: skin papilloma (right foo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to not meeting study endpoints as defined per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT03095248/Prot_SAP_000.pdf